CLINICAL TRIAL: NCT04980053
Title: The Impact of Back and Breast Massage Practised on Mothers With Preterm Birth on the Amount of Milk and Level of Anxiety
Brief Title: The Impact of Back and Breast Massage
Acronym: Massage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seyma Kilci Erciyas (Other)
Responsible Party: Sponsor-Investigator, Seyma Kilci Erciyas, Lecturer, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: Seyma Kilci Erciyas
Record Dates: First submitted 2021-06-20; First posted 2021-07-28 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Premature Birth
Keywords: breast massage; breast milk; back massage; oxytocın; anxıety
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Intervention Model Description: 20 for intervention 1 (back massage) group, 20 for intervention 2 (breast massage) group and 20 for control group
Who Masked: Participant, Outcomes Assessor
Masking Description: In this context, individuals included in the study will be assigned to the control and intervention groups respectively, randomized by an expert statistician and received in closed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Back Massage (Experimental): Back massage will be initiated in the first 2 hours after birth and it will be performed every 6 hours for 15 minutes until the mother is discharged from the hospital. After the mother's outfits are removed and the mother is situated in a suitable position, the back of the mother will be massaged by euphlorage, petrissage, friction methods. Then, the participant"s breast will be milked by hand every 3 hours and will be measured in the breast milk storage bag and delivered to the baby nurses until the 5th-7th day.
  Interventions: Other: massage
- Breast Massage (Experimental): Breast massage will be initiated in the first 2 hours after delivery and it will be practised every 6 hours until being discharged. After the researcher washes her hands, the participant's outfits are removed and she is situated in a sitting position, the massage will be practised on both breasts for 10 minutes by the researcher herself. After the mother's breast will be milked by hand every 3 hours and the milk obtained from the breast will be measured in the breast milk storage bag and delivered to the baby nurses.
  Interventions: Other: massage
- Control Group (No Intervention): No intervention will be made to the control group, standard hospital procedures will be applied and the relevant forms will be filled out. Until the mother is discharged from the hospital, the amount of milk obtained from the mother will be measured every 3 hours by the researcher.

INTERVENTIONS:
Other: massage — Intervention group Control group
  Other Names: back massage; breast massage
  Arms: Back Massage; Breast Massage

SUMMARY:
In the study, selections to the experimental and control groups will be made randomly and simple randomization method will be used. In this context, the individuals included in the research will be assigned to the control and initiative groups respectively and randomized by an expert statistician.The sample of the study was found to be at the 95% confidence interval and at the level of α= 0.05. The effect size was found to be 0.5703 based on previous studies. With a theoretical power of 0.95, the minimum sample size was totally calculated as 51, 17 for the intervention 1 (back massage), 17 for the intervention 2 (breast massage) group and 17 for the control group. However, it was aimed to reach 60 people by predicting that there might be case losses, and it was planned to recruit 20 people for each group.

The dependent variables of the study are the amount of breast milk and the level of anxiety. The independent variable is the back and breast massage practice.

This research will be carried out in Zonguldak Gynecology and Pediatrics Hospital between 1st July 2021-2022.

DETAILED DESCRIPTION:
The data of the research will be collected in two phases. In the first phase, the data will be collected by the researcher by face-to-face interview technique with mothers having just given birth in the hospital and meeting the inclusion criteria of the study. At this phase, "Informed Consent Form" prepared by the researcher in line with the literature, "Personal Information Form", "Breastmilk Evaluation Form" and "State-Trait Anxiety Scale" will be used to collect data.

In addition, a digital thermometer to adjust the room temperature and milk storage bags to store the milk will be used. In the second phase, data will be collected by calling the mothers by phone (audio, video) after they are discharged from the hospital. At this phase, "Post-Discharge Breast Milk Evaluation Form", "State-Trait Anxiety Scale" and "New-born Nutritional Status Evaluation Form" will be used. "Personal Information Form", which will be used in the collection of data consists of 20 questions about the socio-demographic characteristics (age, education level, region of residence until the age of 15, spouse's education level, employment status, occupation, family type, income status), fertility characteristics (number of pregnancies, week of birth, type of birth, the state of oxytocin given at birth, planning status of pregnancy, encountering problems during pregnancy, baby's gender and birth weight, baby's height and head circumference), APGAR score of the baby, the person that make her give birth and mother's body mass index, the status of smoking and medicine or herbal product usage to increase breast milk. Informed consent will be obtained if women meeting the inclusion criteria agree to participate in the research. After obtaining their consent, a pre-test will be applied to the women with the "Personal Information Form" and the "State-Trait Anxiety Scale" by face-to-face interview technique. Both state and trait anxiety scales are of 4-point Likert type. There are 10 reversed statements in the state anxiety scale and 7 reversed statements in the trait anxiety scale. In the state anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. Direct statements express negative emotions, reversed statements express positive emotions. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety. According to Öner, in Spielberg's state and trait anxiety inventory, 0-19 points is evaluated as no anxiety, 20-39 points as mild anxiety, 40-59 points as moderate anxiety, 60-79 points as severe anxiety and 80 points as severe anxiety-panic).

Randomized assignment to the experimental and control groups will be made by a statistician in order to control the randomization and selection bias in the study. Participants will be included in initiative 1 (back massage), initiative 2 (breast massage) or control group according to randomized assignments after pre-test application.

Implementation of the Research in the Control Group No intervention will be made to the control group, standard hospital procedures will be applied and the relevant forms will be filled out. Until the mother is discharged from the hospital, the amount of milk obtained from the mother will be measured by the researcher with the "Breast Milk Evaluation Form", and the breast milk will be measured in the storage bag and delivered to the baby nurses. Covid-19 precautions will be taken in all controls of the mother (hand washing, surgical mask, gloves, apron, face visor). When the mother is discharged from the hospital, the "Post-Discharge Breast Milk Evaluation Form" will be given to the mother and she will be told how to fill it out. The contact numbers of the mothers will be received and information about the measurements filled in the form will be obtained twice a day. Anxiety levels of mothers will be determined with a post-test using the "State-Trait Anxiety Scale", just before their discharge from hospital and on the 5th-7th days. The mothers will be called again at the 6th week of postpartum, and the "New-born Nutritional Status Evaluation Form" will be applied.

Implementation of Research in the Initiative Group The first back massage will be initiated in the first 2 hours after birth and it will be performed every 6 hours for 15 minutes (first 2 hours, 6th, 12th, 18th, 24th, 30th, 36th, 42nd, 48th hour, etc.) until the mother is discharged from the hospital. After the mother's outfits are removed and the mother is situated in a suitable position, the back of the mother will be massaged by euphlorage (stroking), petrissage (pressing the back), friction methods. Then, the mother's breast will be milked by hand and the milk obtained from the breast will be measured in the breast milk storage bag and delivered to the baby nurses. The amount of milk will be measured with the "Breast Milk Evaluation Form".

Before the mother's being discharged from the hospital, a family member will be taught about the fact that how the back massage is practised and asked to practise it at home until the 5th-7th day. The video for the practice of the back massage to be applied at home will be taken by the researcher. Both the video and the brochures will be given to the mother and the person who will apply the massage. Before the mother's being discharged, whether the family member practises the massage correctly or not will be observed. After being discharged, video or audio calls will be made with the family member and asked about whether he/she practices the back massage on the mother and the effectiveness of the massage will be evaluated. The length of the back massage to be practised at home will be for 15 minutes, four times a day (every 6 hours) that is in the morning, at noon, in the evening and at night. Besides this, when the mother is discharged from the hospital, the "Post-Discharge Breast Milk Evaluation Form" will be given to the mother and she will be told how to fill it out. Information about the form will be obtained twice a day by contacting the mother. Anxiety levels will be determined with a post-test using the "State-Trait Anxiety Scale" (Appendix 5) before being discharged and on the 5th-7th days, with. At the 6th week of postpartum, the breastfeeding status of mothers will be evaluated with the "Nutrition Status of the New-born Evaluation Form".

Initiative 2 (breast massage group): The first breast massage will be initiated in the first 2 hours after delivery and it will be practised every 6 hours (first 2 hours, 6th, 12th, 18th, 24th, 30th, 36th, 42nd. , 48th hour) until being discharged. After the researcher washes her hands, the mother's outfits are removed and she is situated in a sitting position, the massage will be practised on both breasts for 10 minutes by the researcher herself. After the breast massage, the mother will be milked by hand and the milk obtained from the mother will be measured in the breast milk storage bag and delivered to the baby nurses. The amount of milk obtained from the mother will be measured with the "Breast Milk Evaluation Form".

The mother will be taught about the breast massage and asked to practise it at home until the 5th-7th day. A video about the self-practice of breast massage will be taken and given to the mother with the brochures. Self-practice of breast massage takes an average of 2-3 minutes and consists of five steps which are pumping the breast, pressing against the rib cage, clockwise or counter-clockwise circular movements, sliding the breast up and down, and back and forth movements. Each step will be performed five times and before each milking time . Whether the mother practices breast massage correctly or not will be evaluated before her being discharged. After being discharged, video or audio calls will be made with the mother and asked about whether she practices the massage herself and the effectiveness of the massage will be evaluated. In addition, while the mother is being discharged from the hospital, the "Post-Discharge Breast Milk Evaluation Form" will be given to the mother and she will be told how to fill it out. Information about the form will be obtained twice a day by contacting the mother. Anxiety levels will be determined with a post-test using the "State-Trait Anxiety Scale", before being discharged and on the 5th-7th days. At the 6th week of postpartum, the breastfeeding status of mothers will be evaluated with the "Nutrition Status of the New-born Evaluation Form".

ELIGIBILITY:
Inclusion criteria for the research are as follows:

* Having a caesarean or vaginal delivery for the first time,
* Giving preterm birth between 32-37 weeks,
* Having only one baby,
* Having a baby with an APGAR score above 4,
* Having the baby in the intensive care unit or being apart from the baby,
* Not having any psychiatric disease,
* Being aged 18 and over and having no communication problems such as seeing, hearing or speaking.

Exclusion criteria from the research are as follows;

* Having a mental and psychological disorder,
* being HIV-infected
* Having a breast surgery before, or having a history of breast cancer,
* Having breast infection,
* Living apart from the husband or being divorced,
* Having lost the baby.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-06 (Estimated); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Amount of Milk | Change from Amount of Milk 7 Days
  measured in the breast milk storage bag (ml)
Level of Anxiety | 1th day
  The trait anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Level of Anxiety | 7th day
  The trait anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Level of Anxiety | 6th week
  The trait anxiety scale, the responses are classified as (1) Not at all, (2) A little, (3) A lot, and (4) Completely; Responses in the trait anxiety scale are classified as (1) almost never, (2) sometimes, (3) often, and (4) almost always. There are two kinds of statements (direct and reversed) in scales. While scoring these statements, those with a score of 1 turn into 4, and those with a score of 4 turn into 1. In direct statements, responses with a value of 4 indicate high anxiety. In reversed statements, responses with a value of 1 indicate high anxiety while those with a value of 4 indicate low anxiety. The scores obtained from both scales range from 20 to 80. The score obtained from the scales constitutes the individual's score to be interpreted at the level of anxiety. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Socio-demographic characteristics of participant | 1th day
  education level
Socio-demographic characteristics of participant | 1th day
  age
Socio-demographic characteristics of participant | 1th day
  region of residence until the age of 15
Socio-demographic characteristics of participant | 1th day
  spouse's education level,
Socio-demographic characteristics of participant | 1th day
  employment status
Socio-demographic characteristics of participant | 1th day
  occupation
Socio-demographic characteristics of participant | 1th day
  family type
Socio-demographic characteristics of participant | 1th day
  income status
Fertility characteristics of partıcipant | 1th day
  number of pregnancies
Fertility characteristics of partıcipant | 1th day
  week of birth
Fertility characteristics of partıcipant | 1th day
  type of birth
Fertility characteristics of partıcipant | 1th day
  the state of oxytocin given at birth
Fertility characteristics of partıcipant | 1th day
  encountering problems during pregnancy
Fertility characteristics of partıcipant | 1th day
  smoking during pregnancy
Fertility characteristics of partıcipant | 1th day
  to take medicine or herbal product usage to increase breast milk
Fertility characteristics of partıcipant | 1th day
  the person that make her give birth
Fertility characteristics of partıcipant | 1th day
  mother's body mass index (kg/m^2)
Fertility characteristics of partıcipant | 1th day
  mother's weight (kg)
Fertility characteristics of partıcipant | 1th day
  mother's weight (cm)
Fertility characteristics of partıcipant | 1th day
  to take vitamin in pregnancy
Fertility characteristics of partıcipant | 1th day
  to take iron preparation in pregnancy
Fertility characteristics of partıcipant | 1th day
  to take breastfeeding education in pregnancy
Characteristics of baby | 1th day
  baby's gender
Characteristics of baby | 1th day
  birth weight
Characteristics of baby | 1th day
  head circumference
Characteristics of baby | 1th day
  APGAR score
Characteristics of baby | 1th day
  reason for hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma K ERCİYAS, Principal Investigator — Ege University
Locations (1):
- Zonguldak Gynecology and Pediatrics Hospital, Zonguldak, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since this is a doctoral thesis, it is planned to be shared after the thesis is published.